CLINICAL TRIAL: NCT06184750
Title: Refining Tamoxifen Dose for Premenopausal Breast Cancer Risk Reduction (RENAISSANCE): A Phase II Single Arm Trial
Brief Title: Finding the Best Tamoxifen Dose for Breast Cancer Risk Reduction in Premenopausal Women, RENAISSANCE Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2023-10628; NCI-2023-10628 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI23-14-01 (Other: Northwestern University); INT23-14-01 (Other: DCP); P30CA060553 (NIH); UG1CA242596 (NIH); UG1CA242609 (NIH); UG1CA242632 (NIH); UG1CA242635 (NIH); UG1CA242643 (NIH)
Record Dates: First submitted 2023-12-27; First posted 2023-12-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Breast Atypical Ductal Hyperplasia; Breast Atypical Lobular Hyperplasia; Breast Carcinoma; Breast Ductal Carcinoma In Situ; Breast Lobular Carcinoma In Situ; Estrogen Receptor-Positive Breast Carcinoma
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms; Breast Carcinoma In Situ | interventions — Biopsy; Specimen Handling; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prevention (tamoxifen) (Experimental): Participants receive tamoxifen 5mg PO QD for 6 months. Participants with aDAR >= 10% on mammogram at 6 months continue receiving tamoxifen 5mg PO QD for 12 months. Participants with aDAR < 10% at 6 months are escalated to receive tamoxifen 10mg PO QD for 6 months. Participants with aDAR >= 10% after 6 months of tamoxifen 10mg continue receiving tamoxifen 10 mg PO QD for 6 months. Participants with aDAR < 10% after 6 months of tamoxifen 10mg are given the option of continuing tamoxifen 10mg or escalating to receive tamoxifen 20mg PO QD for 6 months. Participants undergo mammography and collection of blood samples at screening and on study. Participants may optionally undergo biopsy at screening and on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Mammography; Other: Questionnaire Administration; Drug: Tamoxifen

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Mammography — Undergo mammography
  Other Names: MG
Other: Questionnaire Administration — Ancillary studies
Drug: Tamoxifen — Given PO
  Other Names: TMX

SUMMARY:
This phase II trial evaluates response-guided low-dose tamoxifen for reducing breast density in women who are at higher than average risk for breast cancer. Increasing breast density is a well established risk factor for breast cancer. Tamoxifen is a selective estrogen receptor modulator. It works by blocking the effects of the hormone estrogen in the breast. Tamoxifen has been shown to reduce breast density, even at reduced dosages, and is approved for the prevention of breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate whether the overall proportion of premenopausal tamoxifen responders (defined by absolute dense area reduction on mammogram of > 10%) can be increased through a strategy of within-individual dose escalation among non-responders from 5 mg per day to 10 mg per day.

SECONDARY OBJECTIVES:

I. To assess the association of plasma levels of major tamoxifen metabolites with tamoxifen dose and breast density changes from baseline.

II. To evaluate longitudinal change from baseline in serum biomarkers of tamoxifen response at each dose level: sex hormone binding globulin (SHBG), insulin like growth factor 1 (IGF-1) and C-reactive protein (CRP).

III. To assess the association of baseline dense area (continuous variable) with tamoxifen response.

IV. To evaluate the impact of tamoxifen dose on participant-reported symptoms (Breast Eight Symptom Scale, BESS).

V. To evaluate the impact of tamoxifen dose on adherence to final tamoxifen dose.

EXPLORATORY OBJECTIVES:

I. To evaluate breast tissue-based biomarkers (in research biopsy samples) that associate with tamoxifen response at six months, comparing within-person change in responders and non-responder.

II. To assess the association between single nucleotide polymorphisms that overlap between risk of breast cancer and dense are of breasts; and others that relate to efficiency of tamoxifen metabolism.

III. To evaluate change in breast cancer risk estimates from baseline to 18 months, as assessed by an AI (artificial intelligence) tool and compare changes by dose group.

OUTLINE: This is a within-participant dose-escalation study of tamoxifen.

Participants receive tamoxifen 5mg orally (PO) once daily (QD) for 6 months. Participants with absolute dense area reduction (aDAR) >= 10% on mammogram at 6 months continue receiving tamoxifen 5mg PO QD for 12 months. Participants with aDAR < 10% at 6 months are escalated to receive tamoxifen 10mg PO QD for 6 months. Participants with aDAR >= 10% after 6 months of tamoxifen 10mg continue receiving tamoxifen 10 mg PO QD for 6 months. Participants with aDAR < 10% after 6 months of tamoxifen 10mg are given the option of continuing tamoxifen 10mg or escalating to receive tamoxifen 20mg PO QD for 6 months. Participants undergo mammography and collection of blood samples at screening and on study. Participants may optionally undergo biopsy at screening and on study.

After completion of study intervention, patients are followed up at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women at the time of enrollment defined by any of the following:

  * Age under 50 years and regular menstruation (most recent period within the past 3 months)
  * Age under 50 years and continuous hormonal contraception use and at least one intact ovary
  * Women who are not postmenopausal based on serum hormone levels. Women with estradiol =< 30 pg/mL, follicle-stimulating hormone (FSH) >= 30 IU/mL are eligible
* Women with any of the following:

  * A history of unilateral estrogen receptor (ER) positive ductal carcinoma in situ (DCIS) with local therapy completed (as determined by treating physician recommendation and patient acceptance) at least 1 month prior to study entry. (The untreated breast will be the study breast, for both imaging and optional biopsy)
  * Recent or prior lobular carcinoma in situ (LCIS), or any form of epithelial atypia, flat epithelial (FEA), atypical ductal hyperplasia (ADH), or atypical lobular hyperplasia (ALH)
  * Are risk eligible for preventive medication based on a five-year risk of 1.7% or greater, estimated with a validated model: the National Cancer Institute (NCI) Breast Cancer Risk Assessment Tool, Tyrer-Cusick, Breast Cancer Surveillance Consortium. If the Tyrer-Cuzick model is used a ten-year risk of 3.4% or greater is acceptable
  * Are tamoxifen-eligible by American Society of Clinical Oncology (ASCO) guidelines (>= 2-fold increased risk compared to peer if age >= 45 years, and >= 4-fold increased risk if age < 45 years)
  * A history of mantle radiotherapy
  * A moderate penetrance germline pathogenic variant
* Participants ≥ 18 and ≤ 55 years old will be enrolled. Our trial objectives are not relevant to females under 18 years of age since breast cancer is extraordinarily rare in this age group, and there are no guidelines regarding use of tamoxifen in children, even if know to be at very high risk for breast cancer when older. Because no dosing or adverse event (AE) data are currently available on the use of tamoxifen in participants < 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status must be =< 2 (Karnofsky >= 60%)
* Human immunodeficiency virus (HIV)-infected patients are eligible to participate if they are on effective anti-retroviral therapy with undetectable viral load within the prior 6 months
* Women with evidence of chronic hepatitis B virus (HBV) infection, are also eligible if the HBV viral load is undetectable; they may be on suppressive therapy, if indicated
* Women with a history of hepatitis C virus (HCV) infection are eligible if treated and cured. For those who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Women with herpes simplex virus (HSV) infection are eligible if on chronic or as needed (due to a flare) suppressive antiviral therapy
* Hormonal contraceptive users are eligible and should maintain the same oral contraceptive preparation throughout the duration of the trial. For women who have a levonorgestrel-coated intra-uterine device, removal for medical reasons will be allowed
* The effects of tamoxifen on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because tamoxifen is known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Breast Imaging Reporting and Data System (BIRAD) 1 or 2. If BIRAD 0, follow-up diagnostic imaging must be BIRAD 1 or 2 or cleared clinically with radiology recommendation of return to annual screening
* Women who are factor V leiden carriers and have not had a blood clot are eligible, if approved by their treating physician

Exclusion Criteria:

* BIRADS breast density category A on most recent mammogram
* History of selective estrogen receptor modulator (SERM) use within the past 5 years unless:

  * Use was less than 6 months duration in the past 5 years and not used in the 1 year prior to enrollment OR
  * Use was no greater than 2 months duration in the past 1 year and not used in the 6 months prior to enrollment
* History of invasive breast cancer
* Prior bilateral mastectomy or breast augmentation surgery including breast implants. Prior bilateral excisional surgical biopsy, mastopexy (breast lift) or mammoplasty (breast reduction) is allowed, as long as > 1 year has passed since the procedure
* Women with "mosaic mammographic screening views", i.e., whose larger breast size precludes being imaged within a single mammographic screening view
* Current use of a strong CYP3A4 inducer or a strong CYP2D6 inhibitor unless willing and able to discontinue use and switch to an alternative medication for the duration of participation, under the advice of their physician. If the physician believes the current medication cannot be replaced, the participant will not be eligible
* Current use of Warfarin
* Planning to become pregnant within the next two years. Potential study participants will be questioned about this and excluded if they are planning pregnancy over the next 20 months
* History of thromboembolism, pulmonary embolism, thrombotic stroke, arterial thrombosis of the extremity or deep vein thrombosis. A history of superficial thrombophlebitis is allowed
* History of uterine cancer or atypical uterine hyperplasia with uterus intact
* Participants may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to tamoxifen
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because tamoxifen a category D agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with tamoxifen. Breastfeeding should be discontinued if the mother is treated with tamoxifen
* Women with known gene mutations associated with an increased risk for breast cancer such as BRCA1/2, CDH1, PALB2, PTEN, STK11, or P53
* Current use of sex hormones (estrogen, progesterone, or androgens), unless part of oral contraception pills
* Prior invasive cancer, unless curatively treated, and all treatment was completed > 5 years prior to enrollment

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of women who have a response at any time point | At 6, 12, and 18 months
  Tamoxifen response is defined as absolute dense area reduction (aDAR) of >= 10% on mammogram compared to baseline mammogram. A one sample exact binomial test for one proportion will be used, and the exact two-sided p-value will be reported. Response rate for the entire study population, as well as for the group of women who were dose-escalated, will be estimated and reported with the corresponding 95% confidence interval. Absolute and relative changes in dense area will be estimated using descriptive statistics (e.g., mean and standard deviation, or median and interquartile range), and, as a sensitivity analysis, a paired t-test or the signed rank test will be used to determine whether there was a reduction in dense area. Similar descriptive statistics will be performed in each dose sequence group for both the response rate and dense area changes.

SECONDARY OUTCOMES:
Plasma levels of major tamoxifen (TAM) metabolites | At 6, 12, and 18 months
  Will assess the association of plasma levels of major tamoxifen metabolites with tamoxifen dose and breast density changes from baseline. Metabolite levels will be summarized using standard descriptive statistics at each time point, and change patterns examined using graphical tools for longitudinal data. Will also examine the association of TAM metabolite levels in plasma with aDAR over time using exploratory graphical analyses of aDAR versus (vs.) concurrent metabolite level by time point and dose level. The overall analytic approach to determine whether metabolite levels are associated with aDAR will use linear mixed models.
Longitudinal change in serum biomarkers of tamoxifen response | From baseline up to 18 months
  Will evaluate longitudinal change from baseline in serum biomarkers of tamoxifen response at each dose level: sex hormone binding globulin, insulin like growth factor 1 and C-reactive protein. Biomarker values and changes from baseline will be summarized using standard descriptive statistics at each time point by response status. Differences in baseline levels of these biomarkers between different dose sequence groups will be analyzed using linear regression models with biomarker value as the outcome, and dose cohort as the predictor. Will also use linear mixed models to examine biomarker change patterns over time.
Baseline dense area | Up to 18 months
  Will assess the association of baseline dense area (continuous variable) with tamoxifen response. Will be compared using linear regression models between 5 mg responders and non-responders at 6 months, and between dose sequence groups.
Patient-reported symptoms | At baseline, 6, 12, and 18 months
  Will evaluate the impact of tamoxifen dose on participant-reported symptoms using the Breast Eight Symptom Scale. Will examine patient reported outcome (PRO) patterns over time using graphical tools for longitudinal data, and will use descriptive statistics to summarize PRO values at various time points for groups of patients based on their more recent TAM dose level. Changes in PRO from baseline will be summarized similarly. Linear mixed models will be used.
Adherence to final tamoxifen dose | Up to 18 months
  Will evaluate the impact of tamoxifen dose on adherence to final tamoxifen dose. Adherence will be monitored during monthly participant contacts and by pill count and paper diary at each study visit. Will be summarized using descriptive statistics (mean and standard deviation, or median and interquartile range) for each time point and dose level and will be compared between dose levels at each time point using linear regression models. Adverse events will be summarized during each treatment period (0-6, 6-12 and 12-18 months) and dose level, as well as overall for each dose sequence group.

OTHER OUTCOMES:
Breast tissue-based biomarkers | At 6 months
  Will evaluate breast tissue-based biomarkers and their association with tamoxifen response in participants who consent to the optional research biopsies. Will be compared between 5mg responders vs. non-responders at 6 months using a two-sample t-test or Wilcoxon rank sum test. In addition, logistic regression models may be used to determine the joint association between multiple baseline characteristics and tamoxifen response to 5 mg at 6 months.
Single nucleotide polymorphisms (SNPs) | Up to 18 months
  Will evaluate the association between SNPs that overlap between risk of breast cancer and dense area of breasts. Others that relate to efficiency of tamoxifen metabolism will be explored.
Change in breast cancer risk estimates | From baseline to 18 months
  Will evaluate change in breast cancer risk estimates as assessed by an artificial intelligence tool and compare changes by dose group. Changes will be compared between dose sequence groups using a two-sample t-test. In addition, analysis of covariance models may be fitted with 12-month score as the outcome, and dose group and baseline score as predictors.

CONTACTS AND LOCATIONS:
Overall Officials: Seema A Khan, Principal Investigator — Northwestern University
Locations (11):
- United States (11):
  - University of Arizona Cancer Center - Prevention Research Clinic, Tucson, Arizona
  - Northwestern University, Chicago, Illinois
  - University of Illinois College of Medicine - Chicago, Chicago, Illinois
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Case Western Reserve University, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - M D Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm